CLINICAL TRIAL: NCT05988437
Title: Contribution of the Indoor Environment Medical Advisor in the Management of Fibrosing Hypersensitivity Pneumonitis
Acronym: PHSaDom
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0282
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Hypersensitivity Pneumonitis
Keywords: Fibrosing; indoor environment medical advisor
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypersensitivity pneumonitis (HP) is a diffuse infiltrative pneumonitis (DIP) of immuno-allergic origin, caused by exposure to one or more antigenic substances of organic origin, in genetically predisposed individuals. It can take a fibrosing form, eventually leading to chronic respiratory failure. Diagnosis is based on a combination of clinical, biological, CT scan and histological evidence, and is made during multidisciplinary discussions (MDD) of diffuse interstitial lung disease.

The antigens responsible, of domestic or professional origin, may be micro-organisms, animal proteins or chemical agents. However, the antigen remains unknown in almost 50% of cases. Lack of antigen identification is an independent risk factor for death in patients with fibrosing HP. In fibrosing forms, corticosteroid therapy does not appear to improve functional prognosis, and ninedanib, an antifibrosing treatment offered in progressive forms, only slows functional decline. Identifying the causative antigen is therefore an essential element in the overall management of these patients, with the aim of implementing avoidance measures. A medical exposure questionnaire has been translated into French to help physicians identify the antigen.

The serum precipitin assay is a tool developed to help identify sensitization to an antigen. It is all the more useful when investigations are targeted at the patient's suspected exposure. However, their sensitivity and specificity are variable.

The activity of the indoor environment medical advisor (CMEI) has developed in the care of patients with chronic respiratory or allergic pathologies. Their role is to carry out an audit of the dwelling, take environmental measurements to assess the health risk, inform patients about appropriate eviction measures and, in some cases, refer patients to organizations specializing in home improvement.

The CMEI visits the patient's home. The environmental audit includes a rigorous macroscopic examination and microbiological swabs of visible anomalies. The CMEI can also supplement its analysis with electrostatic dust collectors, which are left in the home for 4 weeks, enabling both qualitative and quantitative characterization of antigens.

To date, no study has prospectively evaluated the contribution of CMEI to antigen identification in patients with fibrosing HP. At the Nantes University Hospital and Angers University Hospital, the environmental audit carried out by the CMEI is an integral part of routine patient management in the event of a HP diagnosis.

The main objective of this study is to measure the diagnostic contribution of the indoor environment medical advisor in the identification of antigens responsible for respiratory pathology in patients with fibrosing HP.

DETAILED DESCRIPTION:
Patients will be prospectively recruited as incidental cases during multidisciplinary discussions of diffuse interstitial lung disease organized on a regular monthly basis between university hospitals, private lung specialists and those practising in outlying hospitals.

Once the patient's non-objection has been collected, a medical self-exposure questionnaire will be completed, and the antigens identified by the questionnaire will be listed (time T1).

As in current practice, the indoor environment medical advisor (CMEI) will then visit the patient's home to carry out an environmental audit, including a macroscopic assessment and swabbing for any abnormalities that might suggest risky antigenic exposure. The results of the swab analysis will be collected along with a number of antigens (T2 time). During this visit, a sensor will be placed in the patient's home for a period of 4 weeks, and the results will be collected after 4 weeks in the home with a number of antigens (time T3).

Following these 3 evaluation times, serum precipitins will be collected according to the antigens identified during the 3 visits.

As part of the patient follow-up, a telephone call by the CMEI at 6 months from the initial environmental audit will assess whether eviction of the identified antigens has been effective. Similarly, at 12 months, the CMEI will make another home visit to assess the rate of eviction of the antigens identified at the initial visit.

In parallel, as part of routine care, a clinical and functional evaluation will be carried out at diagnosis, 6 months and 12 months. A radiological assessment involving a chest CT scan will be performed at diagnosis and at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patient of legal age,
* French-speaking patient,
* Patient with a diagnosis of fibrosing PHS following a multidisciplinary discussion of diffuse interstitial lung disease hypersensitivity pneumonitis .
* Patient who had received an information note presenting the study and who had not expressed opposition to participating in this research.

Exclusion Criteria:

* Opposition of the patient to participate in the study,
* Patient under guardianship, curatorship or safeguard of justice,
* Patients who have moved within the last 12 months, or who plan to move within the next 6 months,
* Patients who have already had a visit from the indoor environment medical advisor.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be prospectively recruited as incidental cases during multidisciplinary discussions of diffuse interstitial lung disease (Diffuse Interstitial Lung Disease) organized on a regular monthly basis between hospital-university centers, private lung specialists and those practising in outlying hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-12 (Estimated); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
To measure the diagnostic contribution of the indoor environment medical advisor in the identification of antigens responsible for respiratory pathology in patients with fibrosing hypersensitivity pneumonitis | 1 month
  Difference in the number of hypersensitivity pneumonitis (HP) risk antigens identified on the one hand by the medical exposure questionnaire and on the other by the indoor environment medical consultant in subjects with HP.

SECONDARY OUTCOMES:
Measure the diagnostic contribution of electrostatic dust sensors in the identification of antigens in patients with fibrosing hypersensitivity pneumonitis | 12 month
Quantify the number of antigens identified using the medical exposure questionnaire, the number of antigens identified by the environment medical advisor, and the number of antigens identified using electrostatic sensors | 1 month
Measure the positivity rate of serum precipitins collected in a manner appropriate to the exposures found | 6 months
Measure the application of eviction advice and the rate of eviction of previously identified antigens 6 months and 12 months after the visit of the environment medical advisor | 12 months
Evaluate the clinical evolution of the patient with fibrosing PHS at 6 months after the environment medical advisor assessment | 6 months
Evaluate the clinical evolution of the patient with fibrosing PHS at 12 months after the environment medical advisor assessment | 12 months
Evaluate the functional evolution of the patient with fibrosing PHS at 6 months after the environment medical advisor assessment | 6 months
Evaluate the functional evolution of the patient with fibrosing PHS at 12 months after the environment medical advisor assessment | 12 months
Evaluate the scanographic evolution of the patient with fibrosing PHS at 6 months after the environment medical advisor assessment | 6 months
Evaluate the scanographic evolution of the patient with fibrosing PHS at 12 months after the environment medical advisor assessment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie DIROU, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, Loire-Atlantique, France